CLINICAL TRIAL: NCT05005962
Title: Prospective Registry for Assessment of Acute Ischemic Stroke Patients Treated With Neurothrombectomy Devices in India
Acronym: PRAAN
Status: Completed | Type: Observational
Sponsor: Medtronic Neurovascular Clinical Affairs (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT20026
Record Dates: First submitted 2021-06-29; First posted 2021-08-16 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Acute Ischemic Stroke
Keywords: Acute Ischemic Stroke; Neurothrombectomy; Revascularization
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Acute ischemic patients suffering with stroke: Acute ischemic patients treated with commercially available neurothrombectomy devices in India. The device can be either a stent retriever or aspiration catheter to treat the stroke as per the labeling indications of the products.
  Interventions: Device: Neurothrombectomy

INTERVENTIONS:
Device: Neurothrombectomy — Neurothrombectomy device will be used to treat patients experiencing the AIS due to large intracranial vessel occlusion within 8 hours of last known well to collect real-world data and to access clinical outcomes associated with the use of these devices.

SUMMARY:
PRAAN is a post-market registry designed to collect real-world data associated with the use of Medtronic market release neurothrombectomy devices in acute ischemic stroke (AIS) patients from India.

DETAILED DESCRIPTION:
The objective of this registry is to access clinical outcomes associated with the use of these device in patients experiencing the AIS due to large intracranial vessel occlusion within 8 hours of last known well.

Real-world evidence per Standard-of-care (SOC) will be generated using Medtronic neurothrombectomy devices approved in India, using on-label indications for use in this post-market clinical follow-up registry.

ELIGIBILITY:
Inclusion Criteria:

1. Subject/subject's legally authorized representative has given Informed Consent according to country regulations, and/or EC requirements
2. Subject is 18 years of age or older
3. Subject has experienced an Acute Ischemic Stroke due to large intracranial vessel occlusion in at least one of the following intracranial vessels: internal carotid artery (ICA), M1 and M2 segments of the middle cerebral artery (MCA), basilar, and vertebral arteries
4. Subject has been or will be treated with a Medtronic market-released neuro thrombectomy device as the initial device used to remove the thrombus
5. Subject is willing to participate in a 90-day follow-up visit
6. Treatment within 24 hours of last known well. For subjects with stroke onset >6 hours:

   * ASPECTS score >5 (per DW-MRI) or >6 (per NCCT)
   * NCCT Core Infarct < 70 ml or MRI DWI with < 70 ml core volume or CTP Ratio of volume of ischemic tissue (penumbra) to infarction of ≥1.8 and an absolute volume of potentially reversible ischemia of ≥15ml
7. Pre-Stroke Modified Rankin Scale (mRS) score ≤1 (immediately) prior to stroke onset
8. Pre-treatment National Institutes of Health Stroke Scale (NIHSS)

   * ≥6 and ≤30 for patients with ≤6 hours of stroke onset.
   * ≥10 and ≤30 for patients with >6 hours of stroke onset.

Exclusion Criteria:

1. Concurrent participation in another mechanical neurothrombectomy device trial or any other clinical trial with an active treatment arm or where the study procedure or treatment might confound the study analysis
2. Patients meeting the contraindication as mentioned in the IFU of devices.
3. Significant mass effect with midline shift

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Up to 200 subjects from 15 sites in India
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-05-21 (Actual)

PRIMARY OUTCOMES:
Performance Evaluation | During the Procedure
  Time to revascularization and revascularization assessment at the end of the procedure using mTICI score
Efficacy Evaluation | Day 7/Discharge after the procedure & 3 month after the procedure
  1. NIHSS at day 7 or discharge, whichever comes first
  2. mRS at discharge or day 7
  3. mRS and NIHSS score at 90 days post index stroke procedure
Safety Evaluation | from index procedure till 3 month after the procedure performed
  Incidence of Neurological Events of Interest, All-cause mortality, Procedure-related AEs, Device-related AEs, and all SAEs

SECONDARY OUTCOMES:
Health Economic analysis of neurothrombectomy procedure in the treatment of patients suffering with ACUTE ISCHEMIC STROKE | At subject discharge after the procedure and 3 month after the procedure
  1. Post-acute discharge disposition: discharge to home or any other facility
  2. Subject disposition at study exit
  3. Cost effectiveness: Evaluation of cost effectiveness of Solitaire and/or React Aspiration catheters family of devices will be performed without a statistical test. Therefore, there is no hypothesis test for this ancillary objective. Cost effectiveness will be calculated using a credible model with inputs from the PRAAN study wherever possible (e.g., age, mortality, quality of life). When direct input from the study is not possible, inputs will be derived from prior clinical evidence, from localized outcomes research (within region of from comparable region), or from expert advisory board input. A separate document will outline the plan for evaluating the cost-effectiveness component. Cost effectiveness will be expressed as incremental cost in local currency per quality adjusted life year gained (QALY).

CONTACTS AND LOCATIONS:
Locations (14):
- India (14):
  - Sterling Hospital, Ahmedabad, Gujarat
  - Artemis Hospital, Gurgaon, Haryana
  - Medanta, Gurgaon, Haryana
  - Yashoda Hospital, Secunderabad, Hyderabad
  - Narayana Hrudayalaya, Bengaluru, Karnataka
  - NIMHANS, Bengaluru, Karnataka
  - Sree Chitra Tirunal Institute for Medical Sciences & Technology, Thiruvananthapuram, Kerala
  - Breach Candy Hospital, Mumbai, Maharashtra
  - HN Reliance, Mumbai, Maharashtra
  - CMC Ludhiana, Ludhiana, Punjab
  - SRMC, Chennai, Tamil Nadu
  - Kovai Medical Center & Hospital, Coimbatore, Tamil Nadu
  - Rabindranath Tagore International Institute of Cardiac Sciences, Kolkata, West Bengal
  - Sir Gangaram Hospital, New Delhi

IPD SHARING:
Plan to Share IPD: No